CLINICAL TRIAL: NCT06734832
Title: A Multicenter, Randomized, Double-blind, Controlled Phase III Clinical Trial on the Efficacy, Safety, and Immunogenicity of the Bivalent Enterovirus Inactivated Vaccine (Vero Cell) in Children Aged 6 to 71 Months.
Brief Title: Efficacy, Safety, and Immunogenicity of the Bivalent Inactivated Enterovirus Vaccine (Vero Cell)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-EV71CA16-3001
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hand, Foot, and Mouth Disease（HFMD)
Keywords: bivalent enterovirus inactivated vaccine; Hand, Foot, and Mouth Disease; EV71; CA16; PHASE Ⅲ; vaccine efficacy; immonogenicity; safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): Bivalent enterovirus inactivated vaccine (Vero cell)
  Interventions: Biological: bivalent enterovirus vaccine (Vero cell), inactivated
- control group (Active Comparator): Enterovirus Type 71 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: Enterovirus Type 71 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: bivalent enterovirus vaccine (Vero cell), inactivated — Two doses are administered with a one-month interval between each dose.
  Arms: trial group
Biological: Enterovirus Type 71 Vaccine (Vero Cell), Inactivated — Two doses are administered with a one-month interval between each dose.
  Arms: control group

SUMMARY:
This multicenter, randomized, double-blind, controlled Phase III clinical trial aims to evaluate the efficacy, safety, and immunogenicity of the bivalent enterovirus-inactivated vaccine (Vero cell) in healthy children aged 6 to 71 months.

The main questions it aims to answer are:

* The primary vaccine efficacy of the investigational vaccine against Hand, Foot, and Mouth Disease（HFMD) caused by CA16 infection compared to the control vaccine.
* The neutralizing antibody levels against EV71 in the trial group are non-inferior to those in the control group after two doses of vaccination.

Researchers will compare the bivalent enterovirus-inactivated vaccine (Vero cell) to the EV71-inactivated vaccine (Vero cell) to prevent HFMD and Herpangina(HA).

Participants will be randomly assigned to the trial group and the control group in a 1:1 ratio to receive two doses of the investigational vaccine or the control EV71 vaccine, with a one-month interval between doses.

DETAILED DESCRIPTION:
This trial employs a multicenter, randomized, double-blind, controlled design. With informed consent, 8000 healthy children participants aged 6 to 71 months will be enrolled, with 4000 participants aged 6 to 23 months and 4000 participants aged 24 to 71 months, maintaining a balanced gender ratio. Among them, 4000 participants aged 6 to 23 months and 3600 participants aged 24 to 71 months have no history of EV71 vaccination, while 400 participants aged 24 to 71 months have a history of EV71 vaccination. All participants will be randomly assigned to the trial and control groups at a 1:1 ratio, receiving two doses of the experimental vaccine or the control EV71 vaccine, with a one-month interval between doses.

Each participant enters the case monitoring period after the first dose, which lasts until the end of two consecutive epidemic seasons. The effective monitoring period begins 14 days after the second dose, with the period before being the monitoring window period. During the case monitoring period, if a participant meets the criteria for a suspected case of enterovirus infection through active follow-up by the researcher or self-reporting by the participant's guardian, a throat swab and/or rectal swab will be collected for RT-PCR nucleic acid testing within three days of the first appearance of symptoms, followed by subsequent follow-up/sampling based on the test results. The protective efficacy of the investigational vaccine will be analyzed based on cases caused by laboratory-confirmed CA16 infections. In addition, enterovirus infection cases collected in this study will be subjected to viral isolation and sequencing analysis to understand their genetic subtypes.

Researchers collect all adverse events (AEs) within 30 minutes after each dose for all participants and serious adverse events (SAEs) from the first vaccination dose to six months after the second dose. Furthermore, any AEs reported by the participant's guardian or known through any other means from the first dose to 30 days after the second dose will be paid attention to, recorded truthfully, and included in the analysis.

A subgroup of 2000 participants will be selected for reactogenicity, including 1000 participants aged 6 to 23 months with no history of EV71 vaccination, 800 participants aged 24 to 71 months with no history of EV71 vaccination, and 200 participants aged 24 to 71 months with a history of EV71 vaccination. For the reactogenicity subgroup, diary cards will be used to collect solicited and unsolicited AEs within 0 to 7 days after each dose, and contact cards will be used to collect AEs from 8 to 30 days after each dose.

A subgroup of 1200 participants from the reactogenicity subgroup will be selected for immunogenicity evaluation, including humoral and cellular immunogenicity subgroups.

The humoral immunogenicity subgroup includes 1160 participants aged 6 to 71 months, with 580 participants aged 6 to 23 months with no history of EV71 vaccination, 380 participants aged 24 to 71 months with no history of EV71 vaccination, and 200 participants aged 24 to 71 months with a history of EV71 vaccination. Venous blood of approximately 3.0ml will be collected from the humoral immunogenicity subgroup before the first dose and at 30 days, 6 months, and 12 months after the second dose.

Serum collected from all participants in the humoral immunogenicity subgroup at the above four time points will be used for neutralizing antibody testing against EV71 and CA16, to evaluate the immunogenicity and duration of immunity against EV71 and CA16. Additionally, the first 100 participants with a history of EV71 vaccination and the first 100 participants without a history of EV71 vaccination from the humoral immunogenicity subgroup will be selected for neutralizing antibody testing against CA10 and CA6 using their serum before the first dose and at 30 days after the second dose; the serum of the remaining 960 participants in the humoral immunogenicity subgroup will be used for neutralizing antibody testing against different serotypes of enteroviruses, including EV71 and CA16, before the first dose and at 30 days after the second dose.

From the humoral immunogenicity subgroup, 50 participants aged less than 12 months with no history of EV71 vaccination will be selected to complete the full vaccination through intramuscular injection on the anterolateral thigh, while the rest of the participants complete the full vaccination through intramuscular injection on the deltoid muscle of the upper arm, for analysis of immunogenicity at different injection sites.

The cellular immunogenicity subgroup will include 40 participants aged 24 to 71 months with no history of EV71 vaccination. Venous blood of approximately 3.0ml will be collected before each dose and on the 14th day after each dose for the detection and analysis of mononuclear cell INF-γ and IL-4 expression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6 to 71 months with no history of EV71 vaccination; or healthy children aged 24 to 71 months who have completed two doses of EV71 vaccine at least 6 months prior.
* Guardians who can understand and voluntarily sign the informed consent form.
* Willing and able to comply with all visit schedules, sample collections, vaccinations, and other research procedures.
* Provide proof of identity documents.

Exclusion Criteria:

* A known history of HFMD/HA.
* Uncontrolled chronic diseases or a history of severe illnesses, including but not limited to cardiovascular diseases, blood disorders, liver or kidney diseases, digestive system diseases, respiratory system diseases, malignant tumors, or a history of major functional organ transplantation.
* Autoimmune diseases, immunodeficiency diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid diseases, asplenia, functional asplenia, and HIV infection).
* Abnormal coagulation function (such as coagulation factor deficiencies, and platelet abnormalities).
* Suffering from/having a history of severe neurological diseases (epilepsy, convulsions, or seizures [excluding a history of febrile seizures]) psychiatric disorders, or a family history of psychiatric disorders.
* Various acute diseases or exacerbations of chronic diseases within the last 3 days, or known or suspected active infections.
* Received a vaccine containing CA16 components.
* Received immunosuppressive or other immunomodulatory treatments for ≥14 days within the past 6 months (prednisone ≥2mg/kg/day, or its equivalent; local or inhaled corticosteroids excluded), cytotoxic therapy, or planning to receive such treatment during the trial.
* Received immunoglobulin or other blood products within the past 6 months, or planning to receive such treatment during the trial.
* Received other investigational drugs or vaccines within the past 30 days, or planning to receive such drugs or vaccines during the trial.
* Received live attenuated vaccines or nucleic acid vaccines within the past 14 days, or subunit or inactivated vaccines within the past 7 days.
* Known allergy to any component of the investigational vaccine (inactivated EV71 virus, inactivated CA16 virus, aluminum hydroxide, sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate, injectable water).
* On the day of the planned vaccination with the trial vaccine, there is a fever, with axillary temperature > 37.0°C before vaccination;
* On the day of the planned vaccination with the trial vaccine, the physical examination is not qualified.
* Skin damage, inflammation, ulcers, rash, or scars at the target injection site that may interfere with vaccination or observation of local reactions.
* According to the investigator's judgment, participants have any other factors that make them unsuitable for participation in the clinical trial.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8000 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the primary vaccine efficacy of the trial vaccine against HFMD caused by CA16 infection compared to the control vaccine. | 1 year
  Evaluate the primary vaccine efficacy of the trial vaccine against HFMD caused by CA16 infection, diagnosed by RT-PCR, in children aged 6 to 71 months (with and without a history of EV71 vaccination) 14 days after full vaccination (based on data from at least 47 cases).
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of HFMD attributable to CA16 infection, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days based on data from at least 47 cases until the end of one epidemic seasons.
Evaluate whether the neutralizing antibody levels against EV71 in the trial group are non-inferior to those in the control group after two doses of vaccination. | 60 days
  Evaluate the seroconversion rate and geometric mean titer (GMT) of EV71 neutralizing antibodies in participants aged 6-71 months without a history of EV71 vaccination and negative for EV71 antibodies before immunization, 30 days after full vaccination.

SECONDARY OUTCOMES:
Evaluate the safety of the trial vaccine. | 6 monthes
  1. Monitor the incidence of adverse events (AEs) within 0-30 days after each dose of the trial vaccine.
  2. Monitor the incidence of adverse reacts (ARs) within 0-30 days after each dose of the trial vaccine.
  3. Monitor the incidence of serious adverse events (SAEs) from the start of vaccination until 6 months after the full vaccination.
Evaluate the long-term vaccine efficacy of the trial vaccine compared to the control vaccine against HFMD caused by CA16 infection | 2 years
  Evaluate the vaccine efficacy against CA16 infection-induced HFMD, confirmed by RT-PCR, in the entire population (including those with and without a history of EV71 vaccination) from 14 days after full immunization until the end of two consecutive epidemic seasons.
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of HFMD attributable to CA16 infection, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days until the end of two epidemic seasons.
Evaluate the long-term vaccine efficacy of the trial vaccine compared to the control vaccine against Herpangina(HA) caused by CA16 infection | 2 years
  Evaluate the vaccine efficacy against HA caused by CA16 infection, confirmed by RT-PCR, in the entire population (including those with and without a history of EV71 vaccination) from 14 days after full immunization until the end of two consecutive epidemic seasons.
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of HA attributable to CA16 infection, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days until the end of two epidemic seasons.
Evaluate the seroconversion rate of the neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, assess the seroconversion rate of neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination.
Evaluate the seropositivity rate of neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, assess the seropositivity rate of neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination.
Evaluate the GMT of the neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, assess the GMT of neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination.
Evaluate the geometric mean increase (GMI) of neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, assess the GMI of neutralizing antibodies against CA16 and EV71 in populations without a history of EV71 vaccination.
Evaluate the vaccine efficacy of the trial vaccine compared to the control vaccine against diseases caused by CA16 infection. | 2 years
  Evaluate the vaccine efficacy against CA16 infection-related diseases (such as HFMD, HA, gastrointestinal diseases, etc.), confirmed by RT-PCR, in the entire population (including those with and without a history of EV71 vaccination) 14 days after full immunization.
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of diseases (such as HFMD, HA, gastrointestinal diseases, etc.) attributable to CA16 infection, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days until the end of two epidemic seasons.
Evaluate the vaccine efficacy of the trial vaccine compared to the control vaccine against severe cases caused by CA16 infection. | 2 years
  Evaluate the vaccine efficacy against severe cases caused by CA16 infection, confirmed by RT-PCR, in the entire population (including those with and without a history of EV71 vaccination) 14 days after full immunization.
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of severe cases attributable to CA16 infection, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days until the end of two epidemic seasons.
Evaluate the vaccine efficacy of the trial vaccine compared to the control vaccine against hospitalization cases caused by CA16 infection. | 2 years
  Evaluate the vaccine efficacy against hospitalization cases caused by CA16 infection, confirmed by RT-PCR, in the entire population (including those with and without a history of EV71 vaccination) 14 days after full immunization.
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of hospitalization cases attributable to CA16 infection, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days until the end of two epidemic seasons.
Evaluate the level of cellular immunity induced by the trial vaccine. | 44 days
  Measure the number of IFN-γ and IL-4 spot-forming cells per 3×10^6 peripheral blood mononuclear cells (PBMCs) from participants aged 24 to 71 months without a history of EV71 vaccination, before each immunization and on the 14th day after each vaccination.
Evaluate the immunological persistence of the trial vaccine via the seropositivity rate of neutralizing antibodies against EV71 and CA16. | 12 monthes
  Evaluate the seropositivity rate of neutralizing antibodies against EV71 and CA16 at 6 months and 12 months after the full vaccination.
Evaluate the immunological persistence of the trial vaccine via the GMT of neutralizing antibodies against EV71 and CA16. | 12 monthes
  Evaluate the GMT of neutralizing antibodies against EV71 and CA16 at 6 months and 12 months after the full vaccination.
Evaluate the seroconversion rate of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, evaluate the seroconversion rate of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination.
Evaluate the seropositivity rate of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, evaluate the seropositivity rate of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination.
Evaluate the GMT of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, evaluate the GMT of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination.
Evaluate the GMI of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination. | 60 days
  On the 30th day after full vaccination, evaluate the GMI of neutralizing antibodies against CA16 and EV71 in populations with a history of EV71 vaccination.
Evaluate the cross-immunogenicity of the trial vaccine against CA6 and CA10 via seroconversion rate of neutralizing antibodies against CA10 and CA6. | 60 days
  On the 30th day after full vaccination, assess the seroconversion rate of neutralizing antibodies against CA10 and CA6.
Evaluate the cross-immunogenicity of the trial vaccine against CA6 and CA10 via seropositivity rate of neutralizing antibodies against CA10 and CA6. | 60 days
  On the 30th day after full vaccination, assess the seropositivity rate of neutralizing antibodies against CA10 and CA6.
Evaluate the cross-immunogenicity of the trial vaccine against CA6 and CA10 via GMT of neutralizing antibodies against CA10 and CA6. | 60 days
  On the 30th day after full vaccination, assess the GMT of neutralizing antibodies against CA10 and CA6.
Evaluate the cross-immunogenicity of the trial vaccine against CA6 and CA10 via GMI of neutralizing antibodies against CA10 and CA6. | 60 days
  On the 30th day after full vaccination, assess the GMI of neutralizing antibodies against CA10 and CA6.
Evaluate the cross-immunogenicity of the trial vaccine against different serotypes of enteroviruses, including EV71 and CA16. | 60 days
  In populations with and without a history of EV71 vaccination, assess the GMT of neutralizing antibodies against different serotypes of enteroviruses, including EV71 and CA16, on the 30th day after full vaccination.
Evaluate the vaccine efficacy of the trial vaccine compared to the control vaccine against infection cases of EV71, CA10, CA6, and other enteroviruses. | 2 years
  Evaluate the vaccine efficacy against EV71, CA10, CA6, and other enterovirus infection cases, confirmed by RT-PCR, in the entire population (including those with and without a history of EV71 vaccination) 14 days after full immunization.
  The vaccine's efficacy will be evaluated by monitoring the annual incidence rate of cases attributable to EV71, CA10, CA6, and other enterovirus infections, as confirmed by reverse transcription polymerase chain reaction (RT-PCR) nucleic acid testing, following complete full immunization for 14 days until the end of two epidemic seasons.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Xiaoqiang, Dr., Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention
Locations (4):
- China (4):
  - Anhui Provincial Center for Disease Control and Prevention, Hefei, Anhui
  - Fujian Provincial Center for Disease Control and Prevention, Fujian
  - Guangdong Provincial Center for Disease Control and Prevention, Guangdong
  - Hubei Provincial Center for Disease Control and Prevention, Hubei

IPD SHARING:
Plan to Share IPD: Undecided